CLINICAL TRIAL: NCT01082107
Title: Solar Disinfection of Drinking Water for Use in Developing Countries or in Emergency Situations
Brief Title: Solar Disinfection of Drinking Water
Acronym: SODISWATER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Council for Scientific and Industrial Research, South Africa (Other Government)
Collaborators: Royal College of Surgeons, Ireland (Other); European Union (Other)
Responsible Party: Martella du Preez Senior Ms, CSIR
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EU 031650
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2009-06

CONDITIONS: Diarrhea; Dysentery (Bloody Diarrhea)
MeSH Terms: conditions — Diarrhea; Dysentery

ARMS (1):
- Solar disinfection of drinking water (Other)
  Interventions: Other: Solar disinfection in transparent containers (plastic bottles)

INTERVENTIONS:
Other: Solar disinfection in transparent containers (plastic bottles) — Participants in the study drink solar disinfected (SODIS) water. Solar disinfected water is water (> 3 L) that has been placed in direct sunlight for 6 hours. Participants are expected to drink SODIS treated water for the duration of the study.

SUMMARY:
SODISWATER is a European Union funded health impact assessment study investigating the effect of sunlight to inactivate microbial pathogens in drinking water. This study was done by observing whether children younger than 5 years old who drink solar disinfected water were healthier than those who did not. Health was measured by how often the children had diarrhoea.

Participants were given plastic bottles to place in the sun, water samples were then collected from these plastic bottles to be analyzed. They were also requested to fill in diarrhea diaries.

TESTABLE RESEARCH HYPOTHESES:

Health Impact Assessment: Children who use solar disinfected water will have:

(a) lower morbidity due to non-bloody diarrhoea and bloody diarrhoea (c) increased growth rates (d) lower mortality (e) increased family productivity (f) decreased care-giver burden (g) increased school attendance

DETAILED DESCRIPTION:
The current evidence base for solar disinfection in the prevention of diarrhoeal disease in children rests on three published studies. All share two significant weaknesses: all were carried out in Kenya, in communities which have very high incidences of diarrhoeal disease and water characterised by high levels of both turbidity and microbial contamination. Furthermore, neither of the studies of diarrhoeal disease distinguished between dysentery (associated with significant risk of mortality) and other sorts of diarrhoea, which carry a far lower risk. The present study will extend the evidence base into communities at lower risk and with higher water quality. Furthermore, by using pictorial diaries, dysentery can be analysed as a specific health endpoint. Diarrhoea will be recorded consistent with the World Health organisation definition: three or more loose or watery stools in a 24-hour period and/or stools containing blood or mucus.

AIM OF THE PROJECT IN RELATION TO HEALTH IMPACT ASSESSMENT STUDIES:

The primary aim of the SODISWATER PROJECT is to demonstrate that SODIS is an appropriate intervention against diarrhoeal and waterborne disease among communities in developing countries and those affected by natural or man-made disasters by conducting multi-centred epidemiologically controlled Health Impact Assessments of the SODIS technique across the African Continent under a variety of social, geographical and climactic conditions.

SCIENTIFIC OBJECTIVES OF SODISWATER IN RELATION TO HEALTH IMPACT ASSESSMENT STUDIES:

1. Assessment of the change in health reasonably attributed to the provision of solar disinfected drinking water at the point of use in four African countries
2. Assessment of the relationship between solar disinfected drinking water and selected health indicators (including morbidity due to non-bloody diarrhoea and dysentery, weight loss, mortality, growth rates, productivity, care-giver burden, and school attendance. Mortality will also be monitored but the sample sizes are of insufficient size to produce detailed information and scaling up, to account for this is not possible due to prohibitive costs).
3. Demonstration of the effectiveness of SODIS at household level.
4. Assessment of gender specific issues.
5. Demonstration of the degree of acceptance/ compliance of SODIS as a disinfection method.

ELIGIBILITY:
Inclusion Criteria:

* Presence of one or more children aged less than 5 years in the household

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2006-10; Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Reduction in dysentery and non-dysentery diarrhoeal disease in children under five years old | Duration of the study
  The method comprises pictorial or smiley diaries that record diarrhoea consistent with the World Health Organisation definition: three or more loose or watery stools in a 24-hour period and/or stools containing blood or mucus.The smiley diary allows a person to note any diarrhoeal episodes themselves on a recording form on a daily basis. The happy face is marked by the parent or carer when the child passes a normal stool. If a loose or watery stool is passed by the child, one of the sad faces is marked, and if the child passes blood or mucus in his or her stools the special box is marked.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin G McGuigan, PhD, Principal Investigator — Royal College of Surgeons, Ireland
Locations (1):
- Council for Scientific and Industrial Research (CSIR), Pretoria, Gauteng, South Africa

REFERENCES:
- [Background] Conroy RM, Elmore-Meegan M, Joyce T, McGuigan KG, Barnes J. Solar disinfection of drinking water and diarrhoea in Maasai children: a controlled field trial. Lancet. 1996 Dec 21-28;348(9043):1695-7. doi: 10.1016/S0140-6736(96)02309-4. PMID 8973432
- [Background] Conroy RM, Meegan ME, Joyce T, McGuigan K, Barnes J. Solar disinfection of water reduces diarrhoeal disease: an update. Arch Dis Child. 1999 Oct;81(4):337-8. doi: 10.1136/adc.81.4.337. PMID 10490440
- [Background] Conroy RM, Meegan ME, Joyce T, McGuigan K, Barnes J. Solar disinfection of drinking water protects against cholera in children under 6 years of age. Arch Dis Child. 2001 Oct;85(4):293-5. doi: 10.1136/adc.85.4.293. PMID 11567937
- [Derived] Du Preez M, Mcguigan KG, Conroy RM. Solar disinfection of drinking water in the prevention of dysentery in South African children aged under 5 years: the role of participant motivation. Environ Sci Technol. 2010 Nov 15;44(22):8744-9. doi: 10.1021/es103328j. PMID 20977257
- See also: Click here for more information on SODISWATER, a research project funded by the European Union (EU) under the 6th Framework Programme (FP6) — http://www.rcsi.ie/sodis/